CLINICAL TRIAL: NCT05303545
Title: Physical Activity in People With Sequelae of Poliomyelitis : a Cross-sectional Study
Brief Title: Physical Activity in People With Sequelae of Poliomyelitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Sante Parasport Connecte Synergies (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-003
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Poliomyelitis
Keywords: Exercise; Disabled persons; Rehabilitation; Cross sectional studies; Social inclusion
MeSH Terms: conditions — Poliomyelitis; Motor Activity; Social Inclusion | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects with poliomyelitis sequelae
  Interventions: Other: standard of care for patients with poliomyelitis sequelae

INTERVENTIONS:
Other: standard of care for patients with poliomyelitis sequelae — clinical examination, radiological, biological and physiological examinations.

SUMMARY:
People with disabilities are less physically active than the general population. At present, the physical activity level of people with poliomyelitis sequelae and their barriers to physical activity are unknown.

The aim of this study is to describe the physical activity level of people with poliomyelitis sequelae and their barriers to physical activity.

DETAILED DESCRIPTION:
This is a cross-sectional, monocentric, cohort study of subjects with poliomyelitis sequelae followed in a Physical Medicine and Rehabilitation Department.

All consecutive eligible outpatient subjects consulting to the Physical Medicine and Rehabilitation Department of our university hospital will be included.

Data will be collected from the patients' medical records, in particular data related to their clinical, radiological, biological and physiological examinations.

It is an ancillary study to the NO-AGING study.

ELIGIBILITY:
Inclusion Criteria:

* Consulting to the Physical Medicine and Rehabilitation Department of our university hospital
* Having poliomyelitis sequelae
* No opposition to be enrolled in the study from the patient
* Affiliation to a social security scheme

Exclusion Criteria:

* Disability that does not allow the completion of questionnaires
* Acute intercurrent medical situation
* Use of electric wheelchair
* Under court protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with poliomyelitis sequelae.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | Baseline
  Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) Questionnaire

SECONDARY OUTCOMES:
Barriers of physical activity | Baseline
  Barriers to Physical Activity Questionnaire for People with Mobility Impairments (BPAQ-MI)

CONTACTS AND LOCATIONS:
Overall Officials: François Genêt, MD-PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France; Vincent T Carpentier, MD-MSc, Study Chair — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France
Locations (1):
- Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, Garches, France

IPD SHARING:
Plan to Share IPD: No